CLINICAL TRIAL: NCT05944133
Title: Health Insurance Instability and Mortality Among Patients Receiving Buprenorphine Treatment for Opioid Use Disorder
Brief Title: Health Insurance Instability and Mortality Among Patients Receiving Bup Tx for OUD
Status: Active, not recruiting | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 3UG1DA040314-08S4 (NIH); CTN-0141 (Other: NIDA)
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use Disorder; Opioid Overdose; Death
Keywords: Health Insurance Instability; Medications for Opioid Use Disorder; Treatment Retention
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients enrolled: Patients who are enrolled on health plans during active MOUD treatment.
  Interventions: Other: No intervention, observational retrospective study
- Patients who disenrolled: Patients who disenrolled from health plans during active MOUD treatment.
  Interventions: Other: No intervention, observational retrospective study

INTERVENTIONS:
Other: No intervention, observational retrospective study — No intervention

SUMMARY:
The goal of this multi-site observational cohort study is to link electronic health records (EHR) with novel data sources to examine insurance instability and its association with all-cause and overdose mortality in adult patients who received medications for opioid use disorder (MOUD). The main objectives of the study are:

* Objective 1. Perform data linkage of a cohort of patients who received MOUD with the National Death Index using a probabilistic algorithm for matching records to ascertain fact and cause of death relative to treatment and insurance status.
* Objective 2: Assess the association of insurance instability and risk of death, including all-cause mortality and drug- and alcohol-related overdose mortality.

DETAILED DESCRIPTION:
Amidst the current opioid epidemic, the incidence of opioid use disorder (OUD) has increased and medication-based treatments for opioid use disorder (MOUD) remain underutilized. While long-term MOUD is generally associated with improved health and mortality outcomes, maintaining continuous health insurance coverage is a significant challenge to sustained treatment access. Patients with OUD are likely susceptible to experiencing insurance instability due to volatile employment and variable eligibility for public insurance, which results in frequent plan changes and critical coverage gaps. The economic crisis associated with the current COVID-19 pandemic may result in greater insurance coverage instability and losses, which would leave patients with OUD even more vulnerable. High-risk care transitions and significant disruption of treatment, including discontinuation of OUD treatment, increases risk of relapse, overdose, and mortality. Further, heightened vulnerability to insurance instability among racial/ethnic minorities may contribute to observed disparities in addiction treatment access and retention. Despite the potential for insurance instability to create significant barriers to OUD treatment continuity, current knowledge regarding its health and mortality impacts is limited due to the challenge of capturing and evaluating patient outcomes after disenrollment from health systems.

To address this knowledge gap, this research study will examine the association of health insurance instability and mortality risk among patients receiving buprenorphine treatment for opioid use disorder in a multi-site cohort study, leveraging data across four diverse health systems in the US.

Findings from the study can inform strategies to ensure treatment continuity and promote well-being for patients vulnerable to insurance instability, from utilizing insurance navigators to establishing standards for bridge prescriptions of MOUD during enrollment transitions, and developing policies to address coverage gaps, such as insurance subsidies for people with OUD using opioid settlement funds. Additionally, as EHR data are increasingly important for pragmatic trials, this study will also advance intervention research by identifying data sources and methods to address bias from loss to follow-up, a common concern across clinical trials.

ELIGIBILITY:
The retrospective cohort study will consist of patients 16 years and older who received MOUD between January 1, 2012, through December 31, 2021, with follow-up through December 31, 2022. Evidence of MOUD will be determined by (1) buprenorphine with or without an OUD diagnosis and (2) naltrexone (injectable extended-release (XR) or oral; oral naltrexone is included because it may be prescribed prior to the transition to XR naltrexone) with an OUD diagnosis from pharmacy dispensing or orders data.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We anticipate a study population of >20,000 patients based on preliminary data. There will be no study exclusion criteria based on gender, race, or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 27257 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | January 1, 2012 - December 31, 2022
  Death and cause-of-death data from the National Death Index (NDI) will serve as the primary data source for outcomes. Outcome will be identified across follow-up from start of treatment and up to one year after disenrollment from the health system.
Drug and alcohol-related overdose mortality | January 1, 2012 - December 31, 2022
  Death and cause-of-death data from the National Death Index (NDI) will serve as the primary data source for outcomes. Outcome will be identified across follow-up from start of treatment and up to one year after disenrollment from the health system.

CONTACTS AND LOCATIONS:
Overall Officials: Anh P Nguyen, PhD, Principal Investigator — Kaiser Permanente; Ingrid A Binswanger, MD, Principal Investigator — Kaiser Permanente; Jason M Glanz, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Colorado, Aurora, Colorado, United States